CLINICAL TRIAL: NCT06004622
Title: Effectiveness of Calgary Family Intervention Model Improving on Uncertainty, Family Functioning, and Resilience in Caregivers of Infants and Toddlers Undergoing Open-heart Surgery.
Brief Title: Effectiveness of Calgary Family Intervention Model in Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 202306120RINA
Record Dates: First submitted 2023-08-09; First posted 2023-08-22 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-07

CONDITIONS: Nursing
Keywords: Calgary family intervention model; caregiver; uncertainty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): The control group receives care according to the standard intensive care unit nursing guidelines.
- experimental group (Experimental): The experimental group, in addition to following the standard guidelines, undergoes two brief therapeutic sessions using the Calgary Family Intervention Model. Each session lasts approximately 20 minutes. Both groups complete three questionnaires during the study period. Furthermore, after the study concludes, the experimental group participates in an interview lasting approximately 15 minutes before returning home.
  Interventions: Other: Calgary Family Intervention Model

INTERVENTIONS:
Other: Calgary Family Intervention Model — under two brief therapeutic sessions using the Calgary Family Intervention Model. Each session lasted about 20 minutes and was conducted by a single researcher to maintain consistency. The scheduling of these sessions took into consideration the physiological and emotional stability of the participants. If any issues or difficulties arose during the course of the sessions, they could be paused. The confidentiality and privacy of the discussion content were ensured. The intervention took place in a dedicated room within the intensive care unit, providing sufficient space and privacy.
  Arms: experimental group

SUMMARY:
Effectiveness of Calgary family intervention model improving on uncertainty, family functioning, and resilience in caregivers of infants and toddlers undergoing open-heart surgery.Research hypothesis is The experimental group of caregivers for infants and toddlers undergoing open-heart surgery showed significant differences in uncertainty, family functioning, and family resilience before surgery, prior to transferring out of the intensive care unit, and before discharge.

DETAILED DESCRIPTION:
Background: For caregivers of infants and toddlers with congenital heart disease, the experience of their young children undergoing open-heart surgery brings about uncertainty, including waiting for the child's recovery, providing care in the intensive care unit, and the possibility of death. These uncertainties can significantly impact the caregivers' physical and mental well-being, as well as their ability to provide subsequent care and nurture for the child. Therefore, it is crucial to implement intervention measures that focus on caring for the caregivers, reducing their sense of uncertainty, and implementing effective nursing strategies to enhance family functioning and resilience.

Purpose: This study aims to investigate the effectiveness of implementing the Calgary Family Intervention Model on caregivers of infants and toddlers undergoing open-heart surgery in terms of reducing their uncertainty, improving family functioning, and enhancing resilience.

Methods: This study adopts a quasi-experimental research design and will be conducted at a medical center in northern Taiwan. A total of 96 caregivers of infants and toddlers undergoing open-heart surgery will be recruited, and a pre- and post-test design will be employed with two groups. The control group will receive routine nursing care, while the experimental group will receive routine nursing care supplemented with the Calgary Family Intervention Model, which encompasses cognitive, emotional, and behavioral domains. The experimental group will participate in two therapeutic sessions: 1. The day after surgery and before visiting the child, and 2. Prior to transferring out of the intensive care unit. Both groups will be assessed using the parental uncertainty perception scale, APGAR family function assessment scale, and the family resilience scale as outcome measures. Data will be collected before surgery, prior to transferring out of the intensive care unit, and before discharge. Interviews will be conducted with the experimental group, and data analysis will involve Generalized Estimating Equations (GEE) for quantitative data and content analysis for qualitative data.

Expected contributions: In future clinical practice, this study aims to provide valuable insights into the use of family nursing intervention for caregivers of infants and toddlers undergoing open-heart surgery, specifically in managing the uncertainties associated with the illness context. Through therapeutic conversations, this intervention can help identify family strengths and resources, thereby serving as an important reference strategy for enhancing family resilience.

ELIGIBILITY:
Inclusion Criteria:

1. Father or mother of infants and toddlers aged from 1 month to 3 years (inclusive) undergoing open-heart surgery.
2. Infants and toddlers diagnosed with congenital heart disease who are undergoing their first open-heart surgery.
3. Caregivers who are proficient in the national or Taiwanese language and have normal cognitive abilities.
4. Caregivers who can read and understand Chinese characters, enabling them to complete the questionnaires.
5. After explanation and reading of the informed consent, caregivers will provide written consent for participation.

Exclusion Criteria:

1. Father or mother of newborns who undergoing open-heart surgery within the first month after birth.
2. Caregivers with mental illness or intellectual disabilities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2024-10-14 (Actual)

PRIMARY OUTCOMES:
parental uncertainty perception scale | one year
  The Chinese questionnaire consists of 30 items, categorized into four domains: Ambiguity, Lack of Clarity, Lack of Information, and Unpredictability. The scoring method is based on the Likert scale, with scores ranging from 1 ("Strongly Disagree") to 5 ("Strongly Agree"). The possible total score ranges from 30 to 150, with the overall score being the sum of individual item scores. A higher total score indicates a greater sense of uncertainty.
APGAR family function assessment scale | one year
  The questionnaire encompasses five subscales: Adaptation, Partnership, Growth, Affection, and Resolve. Each subscale consists of one question. A 3-point scoring system is employed, where "Often" is scored as 2 points, "Sometimes" as 1 point, and "Hardly Ever" as 0 points. The total score ranges from 0 to 10. Scores between 7 and 10 indicate a functional family, scores between 4 and 6 suggest a moderately dysfunctional family, and scores from 0 to 3 denote a severely dysfunctional family. In other words, higher scores reflect better family functionality, demonstrating the family's ability to effectively handle problems and make harmonious decisions.
family resilience scale | one year
  The content of this questionnaire consists of 31 items, categorized into three domains: Belief System, Organizational Patterns, and Family Communication Process. The scoring of the questionnaire utilizes a five-point Likert scale, ranging from a minimum of 1 to a maximum of 5. The scale includes responses of "Strongly Disagree" (1 point), "Disagree" (2 points), "Neutral" (3 points), "Agree" (4 points), and "Strongly Agree" (5 points). The total score range is from 31 to 155 points. Higher scores indicate greater family resilience.

SECONDARY OUTCOMES:
Interview Outline | approximately one year.
  Interview Content Based on the research questions, design four open-ended questions to understand the effectiveness of receiving the second Calgary Family Intervention in terms of uncertainty, family functioning, and family resilience:
  1. Before participating in the intervention, what were your worries and concerns about your child? After receiving the intervention, have these worries changed in terms of their intensity? (Uncertainty)
  2. How was the emotional interaction within your family before the intervention? Did the intervention have any impact on your family dynamics? (Family Functioning)
  3. How did your family approach crises before the intervention? How has your family's confidence in overcoming challenges changed after participating in the intervention? (Family Resilience)
  4. Considering your child's entire hospitalization experience and your participation in this research intervention, do you have any suggestions or thoughts to share?

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Wen Chen, doctor, Study Director — National Yang Ming Chiao Tung University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The illness beliefs model: Advancing practice knowledge about illness beliefs, family healing, and family interventions. — https://doi.org/10.1016/j.apnu.2022.07.014
- See also: Family Functioning and Congenital Heart Disease. — https://doi.org/10.36660/ijcs.20210194
- See also: Family resilience and its association with psychosocial adjustment of children with chronic illness: A latent profile analysis. — https://doi.org/10.1016/j.pedn.2021.02.010
- See also: Risk factors for low cardiac output syndrome in children with congenital heart disease undergoing cardiac surgery: A retrospective cohort study. — https://doi.org/10.1186/s12887-020-1972-y
- See also: Family resilience in the oncology setting: Development of an integrative framework. — https://doi.org/10.3389/fpsyg.2018.00666
- See also: Family-focused public health: Supporting homes and families in policy and practice. — https://doi.org/10.3389/fpubh.2019.00059
- See also: The resilient process of the family after diagnosis of childhood chronic illness: A qualitative meta-synthesis. — https://doi.org/10.1016/j.pedn.2022.07.017
- See also: A randomized clinical trial of the building on family strengths program: An education program for parents of children with chronic health conditions. — https://doi.org/10.1007/s10995-013-1273-2
- See also: Mental health problems in parents of children with congenital heart disease. — https://doi.org/10.3389/fped.2017.00102
- See also: Individualized family-centered developmental care: An essential model to address the unique needs of infants with congenital heart disease. — https://doi.org/10.1097/jcn.0000000000000546
- See also: How should we treat representative neonatal surgical diseases with congenital heart disease? — https://doi.org/10.1007/s00383-022-05178-z
- See also: Home care experience and nursing needs of caregivers of children undergoing congenital heart disease operations: A qualitative descriptive study. — https://doi.org/10.1371/journal.pone.0213154
- See also: Family resilience, parenting styles and psychosocial adjustment of children with chronic illness: A cross-sectional study. — https://doi.org/10.3389/fpsyt.2021.646421
- See also: Resilience and associated factors in mothers of children with congenital heart disease: A cross-sectional study. — https://doi.org/10.30476/ijcbnm.2021.89691.1630
- See also: Effects of the family support and psychoeducation program based on the calgary family intervention model on the coping, psychological distress and psychological resilience levels of the family caregivers of chronic psychiatric patients. — https://doi.org/10.1016/j.apnu.2022.07.014
- See also: Interventions in post-intensive care syndrome-family: A systematic literature review. — https://doi.org/10.1097/CCM.0000000000004450
- See also: Incidence and mortality trend of congenital heart disease at the global, regional, and national level, 1990-2017. — http://doi.org/10.1097/md.0000000000020593
- See also: A novel nesting protocol to decrease readmission and increase patient satisfaction following congenital heart surgery. — http://doi.org/10.1016/j.pedn.2018.07.009